CLINICAL TRIAL: NCT07073170
Title: A Phase 1, Participant- and Investigator-Blind, Placebo-Controlled, Multiple-Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Oral Daily Doses of LY3549492 in Chinese Participants With Type 2 Diabetes Mellitus
Brief Title: A Study of LY3549492 in Chinese Participants With Type 2 Diabetes Mellitus
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 27335; J3H-GH-GZNH (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-07-10; First posted 2025-07-18 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LY3549492 Dose 1 (Experimental): Participants will receive LY3549492 orally
  Interventions: Drug: LY3549492
- LY3549492 Dose 2 (Experimental): Participants will receive LY3549492 orally
  Interventions: Drug: LY3549492
- LY3549492 Dose 3 (Experimental): Participants will receive LY3549492 orally
  Interventions: Drug: LY3549492
- Placebo (Placebo Comparator): Participants will receive Placebo orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3549492 — Administered orally
  Arms: LY3549492 Dose 1; LY3549492 Dose 2; LY3549492 Dose 3
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The main purpose of this study is to investigate LY3549492 in Chinese participants with type 2 diabetes. Participation in the study will last about 18 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Are native Chinese
* Have type 2 diabetes for at least 6 months
* Have been treated with diet and exercise, with or without a stable dose of metformin for at least 3 months
* Have hemoglobin A1c (HbA1c) of at least 7% and no greater than 10%
* Have a body mass index (BMI) of at least 20 milligrams per square meter (kg/m2) and no greater than 40 kg/m2
* Have had a stable body weight for the 3 months prior to screening
* Women must not be of childbearing potential

Exclusion Criteria:

* Have type 1 diabetes or have had an episode of ketoacidosis or hyperosmolar state requiring hospitalization
* Have had an episode of severe hypoglycemia within 6 months or have a history of hypoglycemia unawareness
* Have a clinically significant gastric emptying abnormality
* Have or have a history of pancreatitis
* Have signs and symptoms of liver disease, with the exception of non-alcoholic fatty liver disease
* Have a personal or family history of multiple endocrine neoplasia syndrome type 2 or medullary thyroid carcinoma
* Have an uncontrolled endocrine abnormality
* Have an abnormal blood pressure or pulse rate
* Have a 12-lead electrocardiogram (ECG) abnormality
* Have a significant history within the past 6 months or current evidence of comorbidities capable of altering the absorption, metabolism, or elimination of drugs, or of constituting a risk when taking the study intervention, or of interfering with the interpretation of data

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Events (SAE) Considered by the Investigator to be Related to Study Drug Administration | Baseline through Week 14
  A summary of treatment emergent adverse events (TEAEs), SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module.

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of LY3549492 | Predose through Week 13
PK: Area Under the Concentration Versus Time Curve (AUC) of LY3549492 | Predose through Week 13

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- China (3):
  - Peking University People's Hospital, Beijing
  - West China Hospital of Sichuan University, Chengdu
  - Peking University First Hospital, Dongcheng District

IPD SHARING:
Plan to Share IPD: No